CLINICAL TRIAL: NCT02694653
Title: Preoperative Cesarean Section Intravenous Acetaminophen and Postoperative Pain Control: A Blinded Randomized Placebo-Controlled Trial
Brief Title: Preoperative Cesarean Section Intravenous Acetaminophen and Postoperative Pain Control
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Dr. James Neutens, Dean, Graduate School of Medicine, University of Tennessee Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3890
Record Dates: First submitted 2016-01-21; First posted 2016-02-29 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Complications; Cesarean Section
Keywords: C/section, Acetaminophen
MeSH Terms: interventions — Saline Solution; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Arm (Active Comparator): Acetaminophen 1000 mg in 100 mL normal saline IV administered 30 minutes prior to c/section incision to infuse within 15 minutes
  Interventions: Drug: Acetaminophen
- Placebo Arm (Placebo Comparator): 100 mL normal saline IV administered 30 minutes prior to c/section incision to infuse within 15 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 100 mL of normal saline IV given 30 minutes prior to elective c/section incision vs acetaminophen 1000 mg IV
  Other Names: Normal Saline
  Arms: Placebo Arm
Drug: Acetaminophen — 1000 mg acetaminophen in 100 mL normal saline IV given 30 minutes prior to elective c/section incision vs placebo
  Other Names: Tylenol
  Arms: Drug Arm

SUMMARY:
To evaluate the use of maternal opiates for pain control post cesarean delivery in those patients that received intravenous acetaminophen 1000 mg in 150 mL of normal saline, infused 30 minutes prior to incision compared to placebo. A comparison of post delivery length of stay in both study groups will be evaluated for cost effectiveness of the use of acetaminophen. a secondary purpose is to determine the levels of neonatal acetaminophen in cord blood at the time of delivery, since this has never been studied.

DETAILED DESCRIPTION:
Research Protocol

Preoperative Cesarean Section Intravenous Acetaminophen and Postoperative Pain Control: A Blinded Randomized Placebo-Controlled Trial

Background: To date, there has been no study that has analyzed the use of intravenous acetaminophen given preoperatively in scheduled cesarean deliveries. There have been studies in non-obstetrical surgical procedures that have demonstrated better pain scores and less use of opiates post surgery when administered preoperatively. If these study findings were found to be equally effective post-cesarean delivery, then fewer opiates would be used by the mother. This would benefit better ambulation and less bowel dysfunction by the mother and less effect on the newborn if the mother is breast-feeding. Acetaminophen is one the drugs of choice for analgesia in obstetrics, because it has no known effects on the mother or fetus/newborn. The drug has been found to be safe when given intravenously. Likewise, more patients are found to have therapeutic levels when the drug is given intravenously versus oral administration. Lastly, since patients are NPO prior to scheduled surgery, giving a medication orally is not recommended. Of the prospective blinded studies performed to date, small numbers have been used ranging from 20 to 28 in each arm. Intravenous acetaminophen is already being used preoperatively for scheduled cesarean sections at UT Medical Center Labor & Delivery and the presumption by the nursing staff is that the patients who receive this "do better" post-delivery (with less pain and less need for oral opiates), but without a blinded placebo-controlled trial, this finding cannot be proven or reported.

Specific Aims: The primary aim of this study is to see if maternal opiate use is decreased in the postoperative period for the study group which receives 1 gram of acetaminophen prior to scheduled cesarean section. The secondary aim of this study is to evaluate the length of stay of the mother post-delivery in both the study and placebo groups to see if there are any differences. If found to be significant, this can be analyzed for cost effectiveness. Lastly, pain scores will be evaluated to determine if they improved with preoperative acetaminophen. To date no one has ever studied the cord blood levels of acetaminophen following administration close to delivery, and as such no information on normal acetaminophen levels in the newborn is available.

Enrollment: Enrollment will involve all pregnant patients that enter labor and delivery for a scheduled cesarean delivery once the study is started until a total of 150 are obtained. Enrollment will be determined by the Primary physicians involved in the study, or nurse practitioners/research coordinators or any of the anesthesia or obstetrical residents.

Randomization: The study is a prospective randomized placebo controlled trial. Once patients are consented, an order for the medication will be supplied to the Pharmacy Department. The Pharmacy Department will supply the mediation in a 100 mL bag to be infused over 15 minutes just prior to incision. The Pharmacy will randomly supply these as either a placebo bag of normal saline or the study drug of 1000 mg (1 gram) of intravenous acetaminophen in normal saline. No study personnel from OB/GYN or Anesthesia will have results until the study has been completed. The Pharmacy is responsible for maintaining the blinding of this study

Study Procedure: All eligible pregnant patients (as described above) that are admitted to labor and delivery for a scheduled cesarean delivery will be asked to participate in the study. If they meet inclusion criteria and agree, an approved informed consent form (see attached) will be signed. The goal will be to obtain 150 patients. Once the drug bag is received from Pharmacy, it will be infused over 15 minutes, approximately 30 minutes prior to the incision start time. All patients will receive standard preoperative anesthesia and antibiotics per protocol for pain and prevention of surgical site infection.

At delivery, cord blood will be obtained (the newborn will NOT need a blood draw) and this sample will go the laboratory for an acetaminophen level of the fetus.In order to maintain blinding, all 150 cord blood samples will be sent for testing and results will blindly be reported to the Pharmacy.Pharmacy personnel will also keep cord blood levels. No action by the pharmacy personnel for monitoring of cord blood levels will be necessary, as there are no cord blood therapeutic levels available. This study will seek to discover that information.

Post-delivery, pain and medication assessment scoring per UT Medical Center protocol will be performed by the postoperative/postpartum nurses to assess pain control. Patients are currently monitored by the Pharmacy for acetaminophen levels not to exceed 4000 mg/day and this process will continue per hospital protocol. In order to avoid breaking the blind, all study patients will be treated as if they received preop acetaminophen and will then be switched to a non acetaminophen analgesic if a fifth dose of acetaminophen is required. After the first 100 study patients are enrolled, a preliminary study assessment will be performed to see if any significance in study goals (ie: decreased opiate use, length of stay and improved pain scores) is found since statistical differences were seen in other studies with fewer numbers. This information will be collected through chart review by investigators and research assistants which the IRB has approved. If this data collection on the first 100 study patients is found to be significant, the study will be stopped. However, blinding will be maintained until study completion is determined.

Adverse Event: Adverse events related to this study are minimal because the patient will have an intravenous line placed for the surgery whether or not she consents. In addition, all patients receive preoperative antibiotics prior to the surgical delivery so receiving a medication in this fashion is already being done. Furthermore, obtaining cord blood does not involve any laboratory blood draws on the newborn. (No study has ever evaluated the acetaminophen level in cord blood though levels in the newborn following oral administration have not been higher than the maternal levels. The reports on patient levels in other studies have not been in the toxic range following a single administration of 1000 mg. Therefore, though never studied, it is not expected that the cord blood levels will be above the therapeutic range. The molecular weight of acetaminophen is 151 Daltons with a bioavailability of about 75% and a half-life of 1 to 4 hours. Based on these parameters, the drug would be expected to cross into and out of the fetus fairly easily similar to penicillin, creating a fairly steady state within the mother and fetus.) Although adverse events are not expected in either the mother or neonate, the study investigators will be responsible for monitoring any adverse events should that become necessary. Evaluation of maternal and neonatal liver and kidney function is not necessary as the mother will only receive one dose of acetaminophen, 1000 gms, which is considered a normal adult dose.

Study Withdrawal: Any patient at any time can ask to be withdrawn from the study.

Statistics: A formal power analysis has been completed by Dr. Eric Heidel and 150 study subjects has been shown to be more than adequate for this study.

Confidentiality: All patient material will be kept confidential and all patient-identifying information will be deleted once the pain scores, number of opiates dosages received, the length of stay for each participant, and the cord blood acetaminophen level is recorded. The laboratory results will be sent to the Pharmacy Department until study completion to keep the process blinded since all cord blood samples will be tested.

Follow-up / Record Retention: No patient follow-up will occur since the purpose of this study is to basically determine if this preoperative medication protocol is found to be beneficial in the short term post cesarean section. Record retention of study results will be based on the rules of the peer-review journal that accepts the study for publication.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant having an elective c/section

Exclusion Criteria:

* Acetaminophen allergy
* Hepatitis history
* Liver or kidney disease
* Use of Tylenol within 24 hours
* Use of opiates within 24 hours

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Up to 26 months
  Maximum follow up time for assessment

SECONDARY OUTCOMES:
Milligrams of narcotics given | Up to 26 months
  Maximum follow up time for assessment
Milligrams of Acetaminophen in cord blood | At delivery
  Milligrams of Acetaminophen in cord blood at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Craig V. Towers, MD, Principal Investigator — University of Tennessee Graduate School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
Present at national medical conference and publish in medical journal

REFERENCES:
- [Background] Khalili G, Janghorbani M, Saryazdi H, Emaminejad A. Effect of preemptive and preventive acetaminophen on postoperative pain score: a randomized, double-blind trial of patients undergoing lower extremity surgery. J Clin Anesth. 2013 May;25(3):188-92. doi: 10.1016/j.jclinane.2012.09.004. Epub 2013 Apr 6. PMID 23567482
- [Background] Tsang KS, Page J, Mackenney P. Can intravenous paracetamol reduce opioid use in preoperative hip fracture patients? Orthopedics. 2013 Feb;36(2 Suppl):20-4. doi: 10.3928/01477447-20130122-53. PMID 23379572
- [Background] Needleman SM. Safety of rapid intravenous of infusion acetaminophen. Proc (Bayl Univ Med Cent). 2013 Jul;26(3):235-8. doi: 10.1080/08998280.2013.11928969. PMID 23814378
- [Derived] Towers CV, Shelton S, van Nes J, Gregory E, Liske E, Smalley A, Mobley E, Faircloth B, Fortner KB. Preoperative cesarean delivery intravenous acetaminophen treatment for postoperative pain control: a randomized double-blinded placebo control trial. Am J Obstet Gynecol. 2018 Mar;218(3):353.e1-353.e4. doi: 10.1016/j.ajog.2017.12.203. Epub 2017 Dec 21. PMID 29274831